CLINICAL TRIAL: NCT00951119
Title: The Effect of Device-guided Breathing Exercises on Blood Pressure in Diabetic Patients With Hypertension (Resperate-3) A Randomized, Double-blind Controlled Trial
Brief Title: Device-guided Breathing Exercises on Blood Pressure in Diabetic Patients
Acronym: Reperate3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator, Nanne Kleefstra, Prof. dr. Bilo and N. Kleefstra, Medical Research Foundation, The Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Reperate3
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Hypertension in Type 2 Diabetes
Keywords: type 2 diabetes; hypertension; treatment; non-medical
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- resperate device (Experimental): Resperate© is a device that helps to slow down breathing. This device can measure the breathing patterns through a breathing sensor mounted on the upper abdomen or chest. Furthermore, music-like sound patterns can be composed similar to this breathing pattern, which the patient can hear through the headphones of the Resperate©. By prolonging the expiration, which can be voluntarily used by the user, the frequency of respiration can be slowed down and become more stable (aim"<10 breathings per minute).
  Interventions: Device: Resperate
- control device (Sham Comparator): Resperate device without slowing of breathing
  Interventions: Device: Resperate

INTERVENTIONS:
Device: Resperate — device-guided breathing exercises
  Arms: resperate device
Device: Resperate — breathing device without slowing of breathing frequency
  Arms: control device

SUMMARY:
Rationale: Hypertension is an important risk factor of cardiovascular disease, especially in patients with type 2 diabetes mellitus (T2DM). A relatively recent development for the treatment of hypertension is the use of breathing exercises. The investigators' previous studies with a breathing device did not show any positive results. However, these studies and other trials investigating the effects of breathing devices had not a double-blind design. Therefore, the investigators want to perform a randomized, double-blind, controlled trial in a population of T2DM patients.

Objective: To determine the effect of a device slowing breathing (Resperate©) on office systolic blood pressure (SBP) in diabetic patients with treated hypertension with moderate BP control.

Study design: A randomized, double-blind, controlled trial.

Study population: Patients with type 2 diabetes mellitus, over 18 years old and a baseline systolic blood pressure between 140-160 mm Hg.

Intervention: One group receives treatment with a breathing device (Resperate©) and the other group receives treatment with a "control" breathing device. The latter device does not try to alter the breathing pattern.

Main study parameters/endpoints: The effect of the breathing device on SBP is the main study parameter. Secondary endpoints include diastolic blood pressure (DBP) and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* known T2DM,
* over 18 years old,
* known hypertension with a systolic BP (SBP) between 130-170 mm Hg at the previous visit to the internal outpatient department and at the last visit to the internist (which is the same day as baseline measurement) and treated with one or more anti-hypertensive drugs, which have not been changed for the preceding three months. At baseline the SBP should be between 140-160 mm Hg, measured by the investigator.

Exclusion Criteria:

* patients with orthostatic hypotension,
* known heart failure (NYHA III-IV) and/or patients with pulmonary disease (for example asthma, chronic obstructive pulmonary disease and pulmonary fibrosis),
* patients with insufficient knowledge of the Dutch language to understand the requirements of the study,
* additional criteria were hospitalization in the past 3 months, deafness, blindness and cognitive abilities deemed insufficient for operation of a study device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-09; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The effect of the breathing device on SBP is the main study parameter | 8 weeks

SECONDARY OUTCOMES:
Secondary endpoints include diastolic blood pressure (DBP) and quality of life. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: HEnk J.G. Bilo, MD, PhD, Professor, FRCP, Study Director — Diabetes centre, isala clinics
Locations (2):
- Netherlands (2):
  - Isala Clinics, Diabetes Centre, Zwolle
  - Isala clinics, Zwolle